CLINICAL TRIAL: NCT06493305
Title: The Effect of Neurolingualistik Programming (NLP) on Pain Score, Fear of Pain and Pain Catastrophizing Before Uterine Curettage Due to the Fetal Demise
Brief Title: The Effect of NLP on Pain Before Uterine Curettage Due to the Fetal Demise
Acronym: NLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024- Seah1
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Nursing Caries; Pain, Acute; Pregnancy Loss
Keywords: NLP; uterin curettage; pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Neurolinguistic Programming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No intervention before, after pregnancy termination, pain scores and pain evaluation by questionnaires will be done.
- intervention (Active Comparator): Neurolinguistic programme will be done before uterine curettage for pregnancy termination, after this, pain scores and pain evaluation by questionnaires will be done.
  Interventions: Behavioral: Neurolinguistic programming

INTERVENTIONS:
Behavioral: Neurolinguistic programming — In the NLP application protocol, the visual, auditory and/or tactile representation system that the woman uses most frequently will be determined. Then, using the anchoring technique, the internal reactions and external reactions created by the woman's current symptoms and emotions and thoughts regarding the urination process will be combined using the anchoring technique. Existing negative emotions will be reduced and positive emotions will be reinforced. Then, with the swish technique, the intensity of the woman's existing negative emotions will be erased from the most frequently used visual, auditory or tactile representation system. Then, taking into account the representation system that the woman uses most frequently, the belief change model will be used in her negative thoughts about the current symptom, and her negative feelings and thoughts will be replaced by positive feelings and thoughts and reinforced.
  Arms: intervention

SUMMARY:
Pregnancy termination is a difficult and painful procedure can be done by medically or uterine curettage. Studies have been conducted to reduce the anxiety of women undergoing pregnancy termination, but there are no publications on topics such as anxiety, pain perception, and pain catastrophizing.

Neuro Linguistic Programming (NLP) has been called "the art and science of personal excellence", "the study of subjective experience". NLP helps us understand the difference between our actions that produce mediocre results or failure and those that require success or excellence.

NLP: "How do I do something I do well?", "How can I do it better?", "How can I gain skills that I admire in others? It addresses questions like ". It is important to note that NLP is not limited to observable behavior. Our way of thinking, that is, all experience and it also includes the mental processes that control our actions. By dealing with the entire structure of a person's experience (in fact, their motivation), it tries to shape the thought processes, emotions and beliefs that result in a behavior. It is especially about our communication with ourselves as well as with others.

No study was planned on pain and pain perception during pregnancy termination by uterine curettage by teaching the NLP technique to the patients.

DETAILED DESCRIPTION:
In this randomized controlled study, the group of patients who underwent uterine curettage with the indication of pregnancy termination in the Septic Service of the Department of Gynecology and Obstetrics of Şanlıurfa Training and Research Hospital will be divided into two groups and NLP training will be given before uterine curettage in a double-blind manner and VAS (visual pain scale) after uterine curettage. Evaluation will be made using the fear of pain scale-3 and the pain catastrophizing scale. NLP training will be given for approximately 20 minutes, and the group that will not receive NLP training will remain silent for 20 minutes. The results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, non-pregnant, with an indication for pregnancy termination; Those who agreed to participate in the study, patients who understand and can speak Turkish

Exclusion Criteria:

* Patients who do not meet the inclusion criteria or who have had a previous pregnancy termination

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy termination patients
Enrollment: 100 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
VAS score, pain perception scale and pain catastrophizing scales scores | 1 hour
  pain scale

CONTACTS AND LOCATIONS:
Overall Officials: alev esercan, MD, Study Chair — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
by doi
Supporting Information: Study Protocol
Time Frame: six months

REFERENCES:
- [Derived] Kilicli A, Demir I, Esercan A. Effect of neuro-linguistic programming applied prior to uterine curettage for fetal demise on pain score, fear of pain and pain catastrophizing: Randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2025 Sep;313:114592. doi: 10.1016/j.ejogrb.2025.114592. Epub 2025 Jul 21. PMID 40763452